CLINICAL TRIAL: NCT01127191
Title: Effect of Prolonged Military Exercises With High Load Carriage, on Neuromuscular Fatigue and Physiological/Biomechanical Responses
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0901110; 2009-A01346-51 (Other: AFSSAPS)
Record Dates: First submitted 2010-05-11; First posted 2010-05-20 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: military exercises; neuromuscular fatigue; physiological responses; biomechanical responses; simulated military effort; high load carriage; Healthy voluntary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lactatemia, based on subject's arterialized capillary blood samples analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Military
  Interventions: Other: military equipment

INTERVENTIONS:
Other: military equipment — Military exercise of 24 hours

SUMMARY:
Land military missions generally combine prolonged walking/moderate-pace-running and other physical actions such as creeping, jumping, shooting,… which are associated with the direct carrying of high to severe loads of equipment and supplies (20-30 to 50 kg) by soldiers. For an infantry section, "typical" intervention phases last about 20-24 h and combine variable intensity grades. Consequently, military mission characteristics are an interesting investigation field of human fatigue. Previous studies have investigated human neuromuscular alterations after prolonged "normal" locomotion exercises [Millet et al., 2004, 2009], thus the aim of this study is to characterize the neuromuscular determinants of fatigue induced by a 24-h Simulated Military Effort (SME) and a 4-h Military Road March (MM), both performed with high load carriage. Additionally, the consequences of fatigue on physiological and biomechanical parameters of locomotion will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* to be a male
* to have a VO2max > 45ml/min/kg (mean observed value in military subjects)
* to be aged from 30 to 45
* to be recently retreated from National Army
* to be highly experienced in military efforts
* to be trained in exercises involving load carrying
* to benefit from a social security insurance

Exclusion Criteria:

* All subjects with recent (< 3 month) bone, articular or muscle diseases.
* All subjects presenting a clinic sign of intolerance to testing procedures, especially subjects with knee, ankle, hip or back diseases.
* All subjects intolerant to muddy or wooded environment.
* All subjects presenting a clinic sign of intolerance to exercise, and particularly to running or walking while carrying a load
* All subjects involved at the same time in another medical research
* All subjects militarily active
* All subjects with cardiac or pulmonary identified and known diseases

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: military retreated from national army
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Central fatigue quantification based on voluntary and electrically-induced force measurement on activated muscle. | after a a military exercise of 24 hours
Peripheral fatigue based on electrically-induced force measurement on the same muscle in relaxed condition. | after a a military exercise of 24 hours

SECONDARY OUTCOMES:
Oxygen uptake, carbon-dioxide output, energetic-cost of locomotion and respiratory ratio, based on subject's gas exchanges. | after a a military exercise of 24 hours
Lactatemia, based on subject's arterialized capillary blood samples analysis | after a a military exercise of 24 hours
Muscular electrical activities, based on subject's surface EMG analysis | after a a military exercise of 24 hours
Heart rate frequence | after a a military exercise of 24 hours
Walking and running mechanics, measured by an instrumented treadmill | after a a military exercise of 24 hours
Postural equilibration, measured by a piezo-dynamometric double platform | after a a military exercise of 24 hours
Rate of perceived exertion, measured by the Borg scale ranging from 6 to 20 | after a a military exercise of 24 hours
Perceived comfort, measured by a 10 cm visual analogic scale (VAS) | after a a military exercise of 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Roger OULLION, Dr, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Derived] Grenier JG, Millet GY, Peyrot N, Samozino P, Oullion R, Messonnier L, Morin JB. Effects of extreme-duration heavy load carriage on neuromuscular function and locomotion: a military-based study. PLoS One. 2012;7(8):e43586. doi: 10.1371/journal.pone.0043586. Epub 2012 Aug 22. PMID 22927995